CLINICAL TRIAL: NCT03360734
Title: A Phase Ib Study to Evaluate the Safety, Tolerability and Efficacy of Gatipotuzumab and Tomuzotuximab Combination in Patients With EGFR-Positive Metastatic Solid Tumors
Brief Title: Combination of Gatipotuzumab and Tomuzotuximab in Patients With Solid Tumors
Acronym: GATTO
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Glycotope GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5225101; 2017-001609-33 (EudraCT Number)
Record Dates: First submitted 2017-11-20; First posted 2017-12-04 (Actual); Last update posted 2021-07-12 (Actual); Status verified 2021-07

CONDITIONS: Solid Tumor, Adult
MeSH Terms: interventions — Cetuximab; Panitumumab; necitumumab; PankoMab-GEX; GAT

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Combination (Experimental): First part: Combination of Gatipotuzumab (GAT) and Tomuzotuximab (TOM) Treatment: 5 weeks monotherapy with TOM (Day 1: 60mg, Day 2: 660mg, Week 2: 1200mg, Week 4: 1200mg). Then combination of 1200mg TOM with 1400mg of GAT every two weeks until disease progression, as long as patient does not meet any other discontinuation criterion such as unacceptable toxicity.
  Second part: Combination of GAT and TOM or an approved anti-EGFR antibody, i.e. Cetuximab, Panitumumab, or Necitumumab Treatment: One week monotherapy with TOM (Week 1, Day 1: 60mg, Day 2: 660mg). Then 1200mg TOM in combination with 1400mg of GAT every two weeks until disease progression, as long as patient does not meet any other discontinuation criterion such as unacceptable toxicity or commercial anti-EGFR antibody (dosage according to local practices) in combination with 1400mg of GAT every two weeks until disease progression or until unacceptable toxicity
  Interventions: Drug: First part: Gatipotuzumab and Tomuzotuximab; Second part: Gatipotuzumab and Tomuzotuximab or anti-EGFR antibody (Cetuximab, Panitumumab or Necitumumab)

INTERVENTIONS:
Drug: First part: Gatipotuzumab and Tomuzotuximab; Second part: Gatipotuzumab and Tomuzotuximab or anti-EGFR antibody (Cetuximab, Panitumumab or Necitumumab) — Two monoclonal antibodies, Gatipotuzumab is anti-TAMUC1, Tomuzotuximab is anti-EGFR
  Other Names: PankoMab-GEX (GAT) and CetuGEX (TOM)

SUMMARY:
This was a single arm phase Ib study to evaluate the safety and efficacy of combined Tomuzotuximab and Gatipotuzumab therapy in patients with metastatic solid tumors expressing EGFR for whom no standard treatment is available. Patients who had relapsed following their most recent line of chemotherapy and who met all other entry criteria at Screening were enrolled to receive Tomuzotuximab and Gatipotuzumab in combination.

During the extension phase, instead of Tomuzotuximab a commercially avalaible anti-EGFR antibody, i.e. Cetuximab (including any approved biosimilar), Panitumumab, or Necitumumab could be given to patients with cancers for which their use is approved.

DETAILED DESCRIPTION:
Tomuzotuximab (CetuGEX®) is an improved second-generation anti-epidermal growth factor receptor (EGFR) antibody that specifically binds to EGFR and acts as a competitive antagonist at the EGFR ligand binding site.

Gatipotuzumab (PankoMab-GEX®) is a novel glyco-engineered humanized monoclonal antibody, which recognizes the tumor-specific epitope of mucin-1 (TA-MUC1). Gatipotuzumab targets and binds TA-MUC1 epitopes on the surface of tumor cells, potentially activating the immune system to induce ADCC against TA-MUC1 expressing tumor cells.

Based on compelling preclinical evidence suggesting a complex interaction between EGFR and TA-MUC1 expressed on the tumor cell surface in driving carcinogenesis, this study assessed the tolerability, safety and preliminary activity of targeting EGFR and TA-MUC1 with glycoengineered antibodies.

After the safe treatment of 20 patients and the absence of dose-limiting toxicity (DLT), the combination of the two antibodies was considered safe and was started in the second week of treatment for the additional 30 patients to be enrolled in the extension cohort.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female and age ≥18 years
2. Histologically confirmed locally advanced and/or metastatic solid organ tumor including but not limited to the following histology: Non-Small Cell Lung cancer (NSCLC), Gastrointestinal cancer (GI), Breast cancer (BC), Gynecological cancers (GYN). Date of histology should be not older than 18 months from the start of the screening procedures. Additionally 30 patients will be enrolled in 4 expansion cohorts: 1) refractory metastatic Colorectal cancer (mCRC) patients who have failed prior treatment with standard chemotherapeutics and both anti-VEGF and anti-EGFR antibodies; 2) patients with recurrent and/or metastatic Head and Neck cancers, who have failed prior treatment with a checkpoint inhibitor and at least one line of chemotherapy as appropriate depending on the histology and platinum-elegibility; salivary gland tumors can be enrolled in this cohort after failure of at least one line of chemotherapy; 3) refractory metastatic NonSmall Cell Lung cancer (NSCLC) patients who have failed all standard treatment options including chemotherapy, tyrosine kinase inhibitors and immunotherapy as appropriate depending on the histology and mutational status, 4) refractory metastatic Breast cancer (BC) patients who have failed all standard treatment options including chemotherapy, hormone therapy and anti-human epidermal growth factor receptor 2 [HER2] treatment as appropriate depending on the histology.
3. Patients are required to have a positive EGFR IHC expression (≥25% of tumor cells) as assessed by local laboratory. This condition will not be required anymore in the additional 30 patients of the expansion cohorts
4. Measurable disease according to RECIST 1.1. At least 1 lesion, not previously irradiated, that can be accurately measured at baseline as ≥10 mm in the longest diameter (except lymph nodes which must have a short axis ≥15 mm) with computed tomography (CT) or magnetic resonance imaging (MRI) and that is suitable for accurate repeated measurements as per RECIST 1.1 guidelines
5. Failure of standard therapy or non-availability of standard therapy (patients must have received at least one line of chemotherapy and further standard therapy is not an option at study entry)
6. Prior treatment with any anti-EGFR agent should be completed at least 4 months before start of treatment. This condition will no longer be required in the 30 additional patients of the expansion cohorts.
7. Toxicities, except for alopecia and Grade 2 neuropathy, should be not greater than Grade 1 before start of treatment according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE [v. 4.0])
8. Eastern Cooperative Oncology Group (ECOG) Performance Status ≤1 and estimated life expectancy of ≥3 months
9. Adequate organ function as evidenced by the following:

   1. Bone marrow function: hemoglobin ≥90 g/L; white blood cell (WBC) count ≥3.0 x 109/L; absolute neutrophil count (ANC) ≥1.0 x 109/L; platelet count ≥75 x 109/L
   2. Hepatic function: aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5 x upper limit of normal (ULN) (≤5 x ULN if hepatic metastases present); bilirubin ≤1.5 x ULN; alkaline phosphatase ≤5.0 x ULN
   3. Renal function: creatinine <1.5 x ULN
   4. Cardiologic function: LVEF fraction ≥ 50% assessed by radionuclide angiography (MUGA scan) or Echocardiography
10. Patients of both genders with procreative potential must use effective contraception while enrolled in the study and for at least 6 months (for women) or 16 weeks (for men) after the last study drug infusion
11. Written informed consent obtained prior to conducting any study specific procedures

Exclusion Criteria:

1. First 20 patients: Known activating EGFR mutation. This exclusion criterion will no more apply for the 30 additional patients of the expansion cohorts.
2. Involvement in the planning and/or conduct of the study (applies to both Glycotope staff and/or staff at the study site)
3. Concurrent enrolment in another clinical study, unless it is an observational (noninterventional) clinical study or during the follow-up period of an interventional study
4. Patients institutionalized by official means or court order.
5. Chemotherapy, radiation, or any other anti-cancer therapies, including any investigational agent, within 4 weeks prior start of study treatment
6. Concurrent anti-tumor therapy or concurrent immunotherapy
7. Current or prior use of immunosuppressive medication within 28 days before the first dose of study drug. The following are exceptions to this criterion:

   1. Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra articular injection)
   2. Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent
   3. Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication)
8. Major surgery within 4 weeks prior to entering the study and/or incomplete recovery from surgery or planned major surgery
9. Primary or secondary immune deficiency requiring treatment. Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc.]). The following are exceptions to this criterion:

   1. Patients with vitiligo or alopecia
   2. Patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement
   3. Any chronic skin condition that does not require systemic therapy
   4. Patients without active disease in the last 5 years may be included but only after consultation with the study physician
   5. Patients with celiac disease controlled by diet only
10. Clinically active infections >Grade 2 according to the Common Terminology Criteria for Adverse Events (NCI-CTCAE v. 4.0)
11. Patients with known severe allergy or hypersensitivity to other human monoclonal antibodies or who experienced infusion related reactions or other severe toxicity that required permanent interruption of a prior antibody treatment.
12. Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and TB testing in line with local practice), hepatitis B (known positive HBV surface antigen [HBsAg] result), hepatitis C, or human immunodeficiency virus (positive HIV 1/2 antibodies). Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
13. History of another primary malignancy except for: a. Malignancy treated with curative intent and with no known active disease ≥3 years before the first dose of IMP and of low potential risk for recurrence b. Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease c. Adequately treated carcinoma in situ without evidence of disease d. Localized prostate cancer
14. Uncontrolled medical condition considered as high risk for treatment with an investigational drug including unstable diabetes mellitus, vena-cava-syndrome, or chronic symptomatic respiratory disease
15. Clinical signs of brain metastasis or leptomeningeal involvement
16. Symptomatic congestive heart failure (New York Heart Association [NYHA] Class III or IV), unstable angina pectoris or MI within 6 months prior to enrollment, significant cardiac arrhythmia, history of stroke, or transient ischemic attack within 1 year
17. History of seizures, encephalitis, or multiple sclerosis
18. Active drug abuse or chronic alcoholism
19. Pregnant or breastfeeding
20. Known sensitivity to any component of the drugs used
21. Contraindication to the premedication (H1 and/or H2 receptor antagonists and steroids) or commercial anti-EGFR used in this study
22. Legal incompetence, limited legal competence, or detainment in an institution for official or legal reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-11-02 (Actual); Primary Completion 2020-05-04 (Actual); Study Completion 2020-09-29 (Actual)

PRIMARY OUTCOMES:
Safety: Incidence and Severity of adverse events (AEs) and IRRs | 12 months
  Incidence of adverse events (AEs) and IRRs
Overall tolerability | 12 months
  Standard safety assessments in terms of laboratory evaluations, vital signs, electrocardiogram [ECG], and physical examinations

SECONDARY OUTCOMES:
Efficacy of the combined treatment: Objective response rate (ORR) | 12 months
  Objective response rate (ORR), Progression free Survival and Overall survival
Immunogenicity of combined Treatment: incidence of anti-drug antibodies (ADAs) | 12 months
  incidence of anti-drug antibodies (ADAs)
Pharmacokinetics (PK) of combined Treatment: Concentration | 12 months
  Concentration of Gatipotuzumab and Tomuzotuximab in blood and noncompartmental PK parameters

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian Ochsenreither, Dr. med., Principal Investigator — Charité Benjamin Franklin Comprehensive Cancer Center,Hindenburgdamm 30,12200/12203 Berlin, Germany
Locations (4):
- Germany (2):
  - Glycotope-contracted research facility, Berlin
  - Glycotope-contracted research facility, Hamburg
- Glycotope-contracted research facility, Milan, Italy
- Glycotope-contracted research facility, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ochsenreither S, Fiedler WM, Conte GD, Macchini M, Matos I, Habel B, Ahrens-Fath I, Raspagliesi F, Lorusso D, Keilholz U, Rolling C, Kebenko M, Klinghammer KF, Saavedra O, Baumeister H, Zurlo A, Garralda E. Safety and preliminary activity results of the GATTO study, a phase Ib study combining the anti-TA-MUC1 antibody gatipotuzumab with the anti-EGFR tomuzotuximab in patients with refractory solid tumors. ESMO Open. 2022 Apr;7(2):100447. doi: 10.1016/j.esmoop.2022.100447. Epub 2022 Apr 6. PMID 35397434